CLINICAL TRIAL: NCT07229859
Title: Robotic Surgery Via Bilateral Axillo-breast Approach for Relatively Low-risk Papillary Thyroid Carcinoma With Lateral Cervical Lymph Node Metastasis: a Safe and Effective Cosmetic Procedure in the Context of Prevalent Thyroid Ultrasound Screening
Status: Completed | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RHEC-D-2021-024
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-10

CONDITIONS: Differentiated Thyroid Cancer (DTC); Robotic Assistance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- robotic modified radical neck dissection group
- open modified radical neck dissection group

SUMMARY:
The goal of this observational study is to learn the efficacy, cosmetic effectiveness and safety of robotic modified radical neck dissection in well-selected cases, through direct comparison with conventional open surgery in low-risk papillary thyroid carcinoma with lateral cervical lymph node metastasis. The main questions it aims to answer are:

Does robotic neck dissection provide tumor clearance equivalent to that of the conventional open approach? How does the postoperative complication rate of the robotic technique compare with open surgery? Are patients satisfied with the cosmetic appearance of the wound following robotic neck dissection? Researchers will compare robotic surgery with conventional open surgery to see if it has the same efficacy, cosmetic effectiveness and safety.

Participants' postoperative recovery will be followed up, and they will provide pain scores and rate their cosmetic satisfaction with the wound.

ELIGIBILITY:
Inclusion Criteria:

* (1) PTC with lateral LN metastasis confirmed by fine needle aspiration (FNA) biopsy;
* (2) maximum tumor size < 3 cm;
* (3) without extrathyroidal extension;
* (4) metastatic LNs in unilateral levels II, III, IV and/or V;
* (5) number of suspicious metastatic LNs based on preoperative ultrasonography < 5;
* (6) maximum metastatic LN diameter < 3 cm.

Exclusion Criteria:

* (1) metastatic LNs in level I or VII;
* (2) metastatic LNs fused with each other or fixed in the neck or extra-nodal extension;
* (3) history of neck surgery or radiation therapy;
* (4) extranodal extension;
* (5) the presence of TERT mutation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population came from a single high-volume thyroid center, with all surgeries performed by the same surgeon.
Sampling Method: Probability Sample
Enrollment: 332 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Number of retrieved Lymph nodes | From enrollment to the end of surgical procedure
postoperative complications | From enrollment to the end of treatment at 1 year
  Vocal cord paralysis; hypocalcemia; spinal accessory nerve injury; chyle leakage

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided